CLINICAL TRIAL: NCT01679730
Title: Changes of Microbiota in Irritable Bowel Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH-100126-F
Record Dates: First submitted 2012-08-21; First posted 2012-09-06 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2012-09

CONDITIONS: Mucosa Associated Bacteria in Small Intestine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- irritable bowel syndrome patients

SUMMARY:
To investigate the changes of gastrointestinal microbiota in irritable bowel syndrome patients by hydrogen breath test and molecular-based analysis of microbiota in gastrointestinal tract

ELIGIBILITY:
Inclusion Criteria:

* Case group: 20 to 80 years old irritable bowel syndrome patients
* Control group: 20 to 80 years old healthy subjects

Exclusion Criteria:

* without writtent informed consent
* contraindications for enteroscopy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Irritable bowel syndrome patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
difference in component of microbiota between cases and controls

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

REFERENCES:
- [Derived] Chung CS, Chang PF, Liao CH, Lee TH, Chen Y, Lee YC, Wu MS, Wang HP, Ni YH. Differences of microbiota in small bowel and faeces between irritable bowel syndrome patients and healthy subjects. Scand J Gastroenterol. 2016;51(4):410-9. doi: 10.3109/00365521.2015.1116107. Epub 2015 Nov 23. PMID 26595305